CLINICAL TRIAL: NCT01915693
Title: Palliative Radiotherapy in Addition to Self-expanding Metal Stent for Improving Dysphagia and Survival in Advanced Oesophageal Cancer: ROCS (Radiotherapy After Oesophageal Cancer Stenting) Study.
Brief Title: ROCS (Radiotherapy After Oesophageal Cancer Stenting) Study
Acronym: ROCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lisette Nixon (Other Government)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Senior Trial Manager, Velindre NHS Trust
Organization: Velindre NHS Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCTU030; 10/50/49 (Other Grant/Funding Number: National Institute for Health Research Health Technology Assessment programme.)
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Oesophageal Cancer
Keywords: Radiotherapy; stent; quality of life
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Self-expanding metal stents (SEMS) (Control Arm) (No Intervention): SEMS insertion will be undertaken in accordance with standard local protocols. Covered or partially covered metal stents will be used and the length type and mode of stent placement will be selected by the clinician. Insertion will occur within two weeks of randomisation.
- Arm B: SEMS plus external beam radiotherapy (Intervention Arm) (Experimental): External beam radiotherapy (EBRT) is routinely available at regional cancer centres across the UK. For palliation of dysphagia in oesophageal cancer, a radiotherapy course delivering a tumour absorbed dose of 20Gy in 5 fractions or 30Gy in 10 fractions within 4 weeks of SEMS insertion.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — External beam radiotherapy (EBRT) delivering a tumour absorbed dose of 20Gy in 5 fractions or 30Gy in 10 fractions.
  Arms: Arm B: SEMS plus external beam radiotherapy (Intervention Arm)

SUMMARY:
The single most distressing symptom for more than 70% of patients with oesophageal cancer is difficulty in swallowing (dysphagia) caused by blockage of the gullet by a tumour. This causes severe restrictions on food intake, physical activity, social functioning and overall quality of life. Amongst the more effective treatments for improving swallowing, is the insertion of a metal stent across the blocked part, which then self-expands to open up the gullet (Self Expanding Metal Stent or SEMS). The addition of radiotherapy may help to improve the problems caused by dysphagia and provide an additional survival benefit.

The purpose of this study is to test the impact of adding radiotherapy to SEMS on:

* the length of time swallow remains improved for
* quality of life
* survival

DETAILED DESCRIPTION:
The primary objective of the study is to assess the impact of radiotherapy in addition to self-expanding metal stent (SEMS) placement on time to progression of patient-reported dysphagia in a patient population unable to undergo surgery.

Patients will be eligible to take part in the trial if they have oesophageal cancer, are in need of SEMS because of dysphagia, are aged 16 years or older, have been clinically assessed to be able to receive radiotherapy, have an expected survival of at least 12 weeks and are able to give written informed consent.

496 patients will be randomised to receive either SEMS alone or SEMS with radiotherapy. The radiotherapy will be given as an outpatient either as five treatments (one per day) over one week, or ten treatments over two weeks. Questionnaires will be completed before treatment, and at weeks two and four and then monthly for up to one year to assess quality of life and cost effectiveness. Interviews will be held with trial participants at three time points to explore their experiences while on the trial. Interviews will also be held with patients who do not consent to take part in the trial to explore their reasons for non-consent.

Treatments:

Arm A: Self-expanding metal stents (SEMS) (Control Arm) SEMS insertion will be undertaken in accordance with standard local protocols. Covered or partially covered metal stents will be used and the length type and mode of stent placement will be selected by the clinician. Insertion will occur within two weeks of randomisation.

Arm B: SEMS plus external beam radiotherapy (Intervention Arm) External beam radiotherapy (EBRT) is routinely available at regional cancer centres across the UK. For palliation of dysphagia in oesophageal cancer, a radiotherapy course delivering a tumour absorbed dose of 20Gy in 5 fractions or 30Gy in 10 fractions within 4 weeks of SEMS insertion.

There will also be a qualitative component of the trial will have two aims: i) to explore the feasibility of patients' recruitment to the trial and ii) to explore participants' experience of the trial interventions. It will examine their experience of consent and recruitment including reasons for declining, and examine patients' motivation to accept randomisation to an intervention which may include extra radiotherapy. This is an optional component and will require separate consent. Patients who do not consent to the trial, but who do consent to the qualitative component, will be interviewed about their reasons for not-consenting as soon as possible after the approach to participate.

Trial participants who consent to the qualitative component will be interviewed three times: at weeks one and four to capture initial decision-making thoughts and then after the interventions (week 8) to explore patients' experience of interventions and perceptions of benefit or detriment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of oesophageal carcinoma excluding small cell histology
2. Not suitable for radical treatment (oesophagectomy or radical chemoradiotherapy) either because of patient choice or medical reasons
3. Dysphagia clinically assessed as needing stent as primary treatment of the dysphagia
4. Age 16 years or over
5. Discussion and treatment decision for stent placement made by an upper GI multi-disciplinary team
6. Clinician assessment of ability to attend for radiotherapy
7. Expected survival of at least 12 weeks
8. Written informed consent
9. Patient has completed baseline Quality of Life Questionnaires (please note, as a minimum patients must have completed OG25)

Exclusion Criteria:

1. Histology of small cell carcinoma type
2. Tumour length of greater than 12 cm
3. Tumour growth within 2 cm of the upper oesophageal sphincter
4. Endoscopic treatment of the tumour, other than dilatation, planned in the peri-stent period
5. Presence of a tracheo-oesophageal fistula
6. Presence of a pacemaker in proposed radiotherapy field
7. Previous radiotherapy to the area of the proposed radiotherapy field
8. Planned endoscopic treatment of the tumour (e.g. laser) in the immediate peri-stenting period
9. Female patient who is pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
patient-reported dysphagia | within one year
  Assess the impact of radiotherapy in addition to self-expanding metal stent (SEMS) placement on time to progression of patient-reported dysphagia in a patient population unable to undergo surgery.

SECONDARY OUTCOMES:
quality of life | within one year
  Assess the impact of combination treatment on core components of health related quality of life
overall survival | one year
  Assess the impact of radiotherapy in addition to SEMS placement on overall survival
morbidity | one year
  Measure morbidity associated with the interventions
re-intervention rate | one year
  Measure re-intervention rates
cost | one year
  Assess the cost of the addition of radiotherapy to SEMS placement

CONTACTS AND LOCATIONS:
Locations (17):
- United Kingdom (17):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Doncaster Royal Infirmary, Doncaster, England
  - James Cook University Hospital, Middlesbrough, England
  - George Eliot Hospital, Nuneaton, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Musgrove Park Hospital, Taunton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Weston General Hospital, Weston-super-Mare, England
  - Ninewells Hospital, Dundee, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Adamson D, Blazeby J, Porter C, Hurt C, Griffiths G, Nelson A, Sewell B, Jones M, Svobodova M, Fitzsimmons D, Nixon L, Fitzgibbon J, Thomas S, Millin A, Crosby T, Staffurth J, Byrne A. Palliative radiotherapy combined with stent insertion to reduce recurrent dysphagia in oesophageal cancer patients: the ROCS RCT. Health Technol Assess. 2021 May;25(31):1-144. doi: 10.3310/hta25310. PMID 34042566
- [Derived] Adamson D, Byrne A, Porter C, Blazeby J, Griffiths G, Nelson A, Sewell B, Jones M, Svobodova M, Fitzsimmons D, Nixon L, Fitzgibbon J, Thomas S, Millin A, Crosby T, Staffurth J, Hurt C. Palliative radiotherapy after oesophageal cancer stenting (ROCS): a multicentre, open-label, phase 3 randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Apr;6(4):292-303. doi: 10.1016/S2468-1253(21)00004-2. Epub 2021 Feb 19. PMID 33610215